CLINICAL TRIAL: NCT05385419
Title: Diagnostic Value of Bronchoscopic and Thoracoscopic Frozen Section Biopsies in Patients With Pleuropulmonary Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Badwy, Mahmoud Abdelhakam Badwy, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 457
Record Dates: First submitted 2022-05-16; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Event of Undetermined Intent (Y21-Y33)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients subjected for bronchoscopy or medical thoracoscopy (Other): Bronchoscopic and thoracoscopic biopsies will be sent for both frozen section and permenant paraffin section
  Interventions: Diagnostic Test: Bronchoscopic and thoracoscopic frozen section biopsies

INTERVENTIONS:
Diagnostic Test: Bronchoscopic and thoracoscopic frozen section biopsies — Flexible bronchoscopy for patients with lung endobronchial lesion, the bronchoscopic biopsy will be sent for frozen section and permenant paraffin section Medical thoracoscopy for patients with undiagnosed pleural effusion, the thoracoscopic biopsy will be sent for both frozen section and permenant paraffin section

SUMMARY:
Lung cancer is the second most commonly diagnosed cancer worldwide, after breast cancer, and its incidence continues to grow. Flexible bronchoscopy is the diagnostic tool of choice to diagnose endobronchial malignancies. It allows inspection and biopsy of any endobronchial abnormalities under direct vision. Despite specimens are obtained under direct vision, there is a significant failure rate. This may necessitate repeating bronchoscopy. To guide the bronchoscopist on the quality and quantity of specimens during bronchoscopic biopsies for the diagnosis of lung cancer is rapid on-site evaluation (ROSE) of cytological specimens. Intra-procedural Frozen Section Evaluation (FROSE) of bronchoscopic biopsy specimens is an alternative to ROSE and helps preventing repeated bronchoscopies. Medical thoracoscopy increases the diagnostic yield of MPE as it offers the clinician a "window" for direct visualization and collection of samples from the parietal pleura.The acquracy of frozen section biopsies in pleural tumours is largely undefined. Confirmation of the pleural malignancy can lead to immediate pleurodesis following the pleural inspection and biopsy. To our knowledge limited studies discussed the value of frozen section in both bronchoscopic and thoracoscopic biopsies.

DETAILED DESCRIPTION:
All included patients will be subjected to the following:

* Full medical history and clinical examination.
* Routine investigation: complete blood count, liver function test, kidney function test, coagulation profile and arterial blood gases.
* Imaging:

  * Chest X-ray.
  * Chest Ultrasound to evaluate the amount of pleural effusion and the presence of adhesions.
  * MSCT Chest with contrast.
* Pleural fluid study including serum pleural albumin gradient (SPAG), Pleural fluid PH and pleural fluid cytology.

Flexible Bronchoscopy (PENTAX, EB-1970TK 3.2) will be done after instillation of lidocaine 2% by spray and procedural sedation with midazolam (0.01-0.1mg\kg) with continuous monitoring for O2 saturation, heart rate, blood preesure and respiratory rate throughout the procedure. The bronchoscope will be introduced into the nasal cavity and advanced to the level of the vocal cords. Lidocaine 2% will be instilled through the bronchoscope to the vocal cords and tracheobronchial tree to minimize cough. Assessment of the appearance and movement of the cords will be done. As the bronchoscope is advanced beyond the vocal cords, careful inspection of the entire airway will be done. Biopsies from abnormal endobronchial lesions or mucosal abnormalities will be performed. Any evidence of narrowing or dynamic collapse, will be assessed. The biopsies will be sent for both frozen section and permenant paraffin section. Once sufficient tissue sample is confirmed the procedure will be terminated. Final assessment of the airway will be performed to ensure adequate hemostasis.

Medical thoracoscopy using (Karl Storz Heine optical 6mm, Tübingen Germany) with single-port-of-entry technique will be performed under local anesthesia and conscious sedation using midazolam (0.01-0.1mg\kg) or mepredine (0.9mg\kg). The point of entery will be guided with chest ultrasonography. Vertical incision will be made with the scalpel (usually near the midaxillary line), through the skin and subcutaneous tissue, appropriate to the size of the used trocar, usually of approximately 10 mm, parallel with and in the middle of the selected intercostal space. Then the trocar will be inserted in a corkscrew motion until the sudden release of resistance (after passing the costal pleura) is felt, while holding the handle of the trocar firmly in the palm of the hand, as index finger is extended. Under direct vision with the thoracoscope, introduction of pneumothorax will be performed and all pleural fluid will be removed and the pleural cavity will be inspected. Suspicious areas (irregularities, nodules, hyperemic lesions) will be biopsied through the working channel of the thoracoscope using the forceps biopsy.The biopsies will be sent for both frozen section and permenant paraffin section. Intraprocedual confirmation of malignancy will be followed immediately with pleurodesis. An intercostal drain will be placed with underwater seal drainage to drain residual air and fluid from the pleural cavity, allowing the lung to re -expand. The indications for removal of chest tubes will be absence of air leakage and cessation of fluid flow (100-150 mL daily).

The specimen prepared for frozen section will be placed on a metal tissue disc which is then secured in a chuck and frozen rapidly to about -20 to -30 °C. The specimen will be embedded in a gel like medium called optimal cutting temperature compound (OCT) and consisting of polyethylene glycol and polyvinyl alcohol. Subsequently it will be cut frozen with the microtome portion of the cryostat, the section will be picked up on a glass slide and stained (usually with hematoxylin and eosin, the H&E stain).

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with suspected lung neoplastic lesion indicated for bronchoscopy -
* Patients presented with undiagnosed pleural effusion (suspected malignant pleural effusion) who are candidate for thoracoscopy

Exclusion Criteria:

* Age <18 years old.
* Contraindications for bronchoscopy:

  * Uncorrectable hypoxemia
  * Unstable angina
  * Uncontrolled arrhythmias
  * Unexplained or severe hypercarbia
  * Uncontrolled asthma
  * Uncorrectable coagulopathy
* Contraindications for thoracoscopy:

  * Transudative pleural effusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
determining the spceficity and sensitivity of bronhcoscopic and thoracoscopic frozen section biopsy | 4 days
  The accuracy of bronchoscopic and thoracoscopic frozen section to be malignant or non malignant or suspicious

REFERENCES:
- [Background] Fielding D, Hopkins P, Serisier D. Frozen section of pleural biopsies at medical thoracoscopy assists in correctly identifying benign disease. Respirology. 2005 Nov;10(5):636-42. doi: 10.1111/j.1440-1843.2005.00761.x. PMID 16268918